CLINICAL TRIAL: NCT02951845
Title: An Exploratory Open-Label, Single Dose, Randomized, Three-Way Crossover Study In Healthy Subjects to Investigate the Food Effect and Oral Bioavailability of Tablet Formulations Relative to Suspension Formulation of JNJ-54416076
Brief Title: Study to Investigate the Food Effect and Oral Bioavailability of Tablet Formulations Relative to Suspension Formulation of JNJ-54416076 in Healthy Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: JNJ-54416076 program has been stopped for strategic business reasons.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR108239; 54416076EDI1002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-10-31; First posted 2016-11-01 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (12):
- Part 1: Treatment Sequence A1B1C1 (Experimental): Participants in Part 1 will only receive single dose of Treatment A1 oral Suspension (25 milligram [mg], Fasted) then Treatment B1 (Direct Compression Tablets, 5*5 mg Tablets, Fasted) followed by Treatment C1 (Direct Compression Tablets (5*5 mg Tablets, Fed) on Day 1 of the treatment period (Days 1 to 4). Successive treatment periods will be separated by a washout period of 14 days (+/- 1 day).
  Interventions: Drug: JNJ-54416076 (Oral Suspension); Drug: JNJ-54416076 (Formulation 1: Direct Compression Tablets)
- Part 1: Treatment Sequence B1C1A1 (Experimental): Participants in Part 1 will only receive single dose of Treatment B1 then Treatment C1 followed by Treatment A1 on Day 1 of the treatment period (Days 1 to 4). Successive treatment periods will be separated by a washout period of 14 days (+/- 1 day).
  Interventions: Drug: JNJ-54416076 (Oral Suspension); Drug: JNJ-54416076 (Formulation 1: Direct Compression Tablets)
- Part 1: Treatment Sequence C1A1B1 (Experimental): Participants in Part 1 will only receive single dose of Treatment C1 then Treatment A1 followed by Treatment B1 on Day 1 of the treatment period (Days 1 to 4). Successive treatment periods will be separated by a washout period of 14 days (+/- 1 day).
  Interventions: Drug: JNJ-54416076 (Oral Suspension); Drug: JNJ-54416076 (Formulation 1: Direct Compression Tablets)
- Part 1: Treatment Sequence A1C1B1 (Experimental): Participants in Part 1 will only receive single dose of Treatment A1 then Treatment C1 followed by Treatment B1 on Day 1 of the treatment period (Days 1 to 4). Successive treatment periods will be separated by a washout period of 14 days (+/- 1 day).
  Interventions: Drug: JNJ-54416076 (Oral Suspension); Drug: JNJ-54416076 (Formulation 1: Direct Compression Tablets)
- Part 1: Treatment Sequence B1A1C1 (Experimental): Participants in Part 1 will only receive single dose of Treatment B1 then Treatment A1 followed by Treatment C1 on Day 1 of the treatment period (Days 1 to 4). Successive treatment periods will be separated by a washout period of 14 days (+/- 1 day).
  Interventions: Drug: JNJ-54416076 (Oral Suspension); Drug: JNJ-54416076 (Formulation 1: Direct Compression Tablets)
- Part 1: Treatment Sequence C1B1A1 (Experimental): Participants in Part 1 will only receive single dose of Treatment C1 then Treatment B1 followed by Treatment A1 on Day 1 of the treatment period (Days 1 to 4). Successive treatment periods will be separated by a washout period of 14 days (+/- 1 day).
  Interventions: Drug: JNJ-54416076 (Oral Suspension); Drug: JNJ-54416076 (Formulation 1: Direct Compression Tablets)
- Part 2: Treatment Sequence A2B2C2 (Experimental): Participants in Part 2 will only receive single dose of Treatment A2 oral Suspension (25 mg, Fasted) then Treatment B2 (Fluid Bed Granulation Tablets (5*5 mg Tablets, Fasted) followed by Treatment C2 (Fluid Bed Granulation Tablets, 5*5 mg Tablets, Fed) on Day 1 of the treatment period (Days 1 to 4). Successive treatment periods will be separated by a washout period of 14 days (+/- 1 day).
  Interventions: Drug: JNJ-54416076 (Oral Suspension); Drug: JNJ-54416076 (Formulation 2: Fluid Bed Granulation Tablets)
- Part 2: Treatment Sequence B2C2A2 (Experimental): Participants in Part 2 will only receive single dose of Treatment B2 then Treatment C2 followed by Treatment A2 on Day 1 of the treatment period (Days 1 to 4). Successive treatment periods will be separated by a washout period of 14 days (+/- 1 day).
  Interventions: Drug: JNJ-54416076 (Oral Suspension); Drug: JNJ-54416076 (Formulation 2: Fluid Bed Granulation Tablets)
- Part 2: Treatment Sequence C2A2B2 (Experimental): Participants in Part 2 will only receive single dose of Treatment C2 then Treatment A2 followed by Treatment B2 on Day 1 of the treatment period (Days 1 to 4). Successive treatment periods will be separated by a washout period of 14 days (+/- 1 day).
  Interventions: Drug: JNJ-54416076 (Oral Suspension); Drug: JNJ-54416076 (Formulation 2: Fluid Bed Granulation Tablets)
- Part 2: Treatment Sequence A2C2B2 (Experimental): Participants in Part 2 will only receive single dose of Treatment A2 then Treatment C2 followed by Treatment B2 on Day 1 of the treatment period (Days 1 to 4). Successive treatment periods will be separated by a washout period of 14 days (+/- 1 day).
  Interventions: Drug: JNJ-54416076 (Oral Suspension); Drug: JNJ-54416076 (Formulation 2: Fluid Bed Granulation Tablets)
- Part 2: Treatment Sequence B2A2C2 (Experimental): Participants in Part 2 will only receive single dose of Treatment B2 then Treatment A2 followed by Treatment C2 on Day 1 of the treatment period (Days 1 to 4). Successive treatment periods will be separated by a washout period of 14 days (+/- 1 day).
  Interventions: Drug: JNJ-54416076 (Oral Suspension); Drug: JNJ-54416076 (Formulation 2: Fluid Bed Granulation Tablets)
- Part 2: Treatment Sequence C2B2A2 (Experimental): Participants in Part 2 will only receive single dose of Treatment C2 then Treatment B2 followed by Treatment A2 on Day 1 of the treatment period (Days 1 to 4). Successive treatment periods will be separated by a washout period of 14 days (+/- 1 day).
  Interventions: Drug: JNJ-54416076 (Oral Suspension); Drug: JNJ-54416076 (Formulation 2: Fluid Bed Granulation Tablets)

INTERVENTIONS:
Drug: JNJ-54416076 (Oral Suspension) — Participants will receive (25 mg) oral suspension of JNJ-54416076 in Part 1 and Part 2.
Drug: JNJ-54416076 (Formulation 1: Direct Compression Tablets) — Participants will receive JNJ-54416076 Tablet formulation 1 (5*5 mg Tablets [25 mg total]) under fasted and fed condition in Part 1.
  Arms: Part 1: Treatment Sequence A1B1C1; Part 1: Treatment Sequence A1C1B1; Part 1: Treatment Sequence B1A1C1; Part 1: Treatment Sequence B1C1A1; Part 1: Treatment Sequence C1A1B1; Part 1: Treatment Sequence C1B1A1
Drug: JNJ-54416076 (Formulation 2: Fluid Bed Granulation Tablets) — Participants will receive JNJ-54416076 Tablet formulation 2 (5*5 mg Tablets [25 mg total]) under fasted and fed condition in Part 2.
  Arms: Part 2: Treatment Sequence A2B2C2; Part 2: Treatment Sequence A2C2B2; Part 2: Treatment Sequence B2A2C2; Part 2: Treatment Sequence B2C2A2; Part 2: Treatment Sequence C2A2B2; Part 2: Treatment Sequence C2B2A2

SUMMARY:
The purpose of the study is to assess the oral bioavailability of the two tablet formulations of JNJ-54416076 relative to the suspension formulation and to investigate the effect of a high fat meal on the pharmacokinetics of the tablet formulation in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Before randomization, a woman must be: 1) Postmenopausal, defined as a) Greater than (>) 45 years of age with amenorrhea for greater than or equal to (>=)18 months, or b) > 45 years of age with amenorrhea for at least 6 months and lesser than (<)18 months and a serum follicle stimulating hormone (FSH) level >40 International units per liter (IU/L), or 2) Surgically sterile due to a hysterectomy, or bilateral oophorectomy, or bilateral tubal occlusion/ligation procedures, and 3) All women must have a negative serum pregnancy test at Screening; and on Day -1 at each treatment period
* Men (including those who have had vasectomies) must agree to use condoms even if their partner is pregnant (this is to ensure that the fetus is not exposed to the study drug through vaginal absorption) and to not donate sperm during the study and for 3 months after receiving the last dose of study drug. Male participants should encourage their female partner to use an effective method (for example (eg), prescription oral contraceptives, contraceptive injections, intrauterine device, and contraceptive patch) of contraception in addition to the condom used by the male study participant
* Healthy on the basis of physical examination, medical history, vital signs, clinical laboratory tests, and 12-lead electrocardiograms (ECGs) performed. If any of the results are abnormal, the participant may be included only if the investigator judges that the abnormalities or deviations from normal are not clinically significant except for liver function and hematology tests. This determination must be recorded in the participant's source documents and initialed by the investigator
* Body Mass Index (BMI) between 18.5 and 29.9 kilogram per square meter (kg/m^2)(inclusive) and body weight >= 50 kilograms
* Blood pressure (after the participant is sitting for 5 minutes) between 90 and 140 millimeter of mercury (mmHg) systolic, inclusive, and between 50 and 90 mmHg diastolic, inclusive at Screening and on Days -2 and -1 of Period 1. If blood pressure is out of range, up to 2 repeated assessments are permitted

Exclusion Criteria:

* History of, or currently active, significant illness or medical disorders, including (but not limited to) cardiovascular disease (including cardiac arrhythmias, myocardial infarction, stroke, peripheral vascular disease), endocrine or metabolic disease (eg, hyper/hypo-thyroidism), hematological disease (eg, von Willebrand's disease or other bleeding disorders), respiratory disease, hepatic or gastrointestinal disease, neurological or psychiatric disease, ophthalmologic disorders (including retinal disorders or cataracts), neoplastic disease, skin disorder, renal disorder, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* History of Gilbert's disease, Dubin-Johnson or Rotor syndrome, or any family history of liver or gallbladder disease that may suggest an underlying genetic disorder
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma-glutamyltransferase (GGT), bilirubin levels (indirect, or direct), or alkaline phosphatase above the upper limit of normal (ULN) of the clinical laboratory's reference range at Screening or at Day -1 of Period 1
* Hemoglobin, hematocrit, or red blood cell count below the lower limit of normal of the clinical laboratory's reference range at Screening. On Day -1 of Period 1, if participants have hemoglobin, hematocrit, or red blood cell count below the lower limit of normal of the laboratory's reference range, the participants may be included if the investigator judges that the abnormalities or deviations from the reference are not clinically significant
* History of cholecystectomy or gallbladder disease
* Known allergies, hypersensitivity, or intolerance to any of the excipients of the formulation
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (for example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11-22 (Actual); Primary Completion 2017-02-17 (Estimated); Study Completion 2017-02-17 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Analyte Concentration (Cmax) | Predose up to Day 4
  Cmax is the maximum observed analyte concentration.
Time to Reach Maximum Concentration (Tmax) | Predose up to Day 4
  Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area Under Concentration Curve from time zero to the last quantifiable (AUC [0-last]) | Predose up to Day 4
  Area under the concentration-time curve (AUC) from time 0 to the time of the last measurable (non-below quantification limit [non-BQL]) concentration, calculated by linear trapezoidal summation.
Area Under the Plasma Concentration Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | Predose up to Day 4
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time calculated as the sum of AUC (0-last) and C (0-last)/lambda(z); wherein AUC (0-last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(0-last) is the last observed quantifiable concentration, and lambda (z) is elimination rate constant.
Apparent Terminal Elimination Half-life (t1/2term) | Predose up to Day 4
  The elimination halflife (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration time curve and calculated as 0.693/apparent terminal elimination rate constant (lambda[z]).

SECONDARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | 5 to 7 days after discharge (Follow-Up Phase )

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Tempe, Arizona, United States